CLINICAL TRIAL: NCT04280354
Title: Prospective Study to Discover New Biomarkers for Early Detection of Sepsis and Prediction of Sepsis-related Mortality in Patients With Severe Community Acquired Pneumonia (sCAP)
Brief Title: Molecular Biomarkers for Sepsis
Status: Terminated | Type: Observational
Why Stopped: Recruitment failure
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Personalized Health Network (SPHN) (Unknown); Personalized Health and Related Technologies (PHRT) initiative of ETH Zürich (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-00297;qu18Egli3
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Severe Community-acquired Pneumonia (sCAP); Infection, Bacterial
Keywords: Community-acquired Pneumonia; biomarker; clinical data warehouse (CDWH); machine learning; data-driven algorithms; multi-dimensional modelling; sepsis-related mortality; Streptococcus pneumoniae
MeSH Terms: conditions — Sepsis; Community-Acquired Pneumonia; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples will be stored in a biobank on sepsis. In particular serum and DNA samples of hosts will be stored for at least 10 years to answer subsequent research questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with severe community acquired pneumonia (cases): Cases: Patients with severe community acquired pneumonia with required ICU admission.
  Interventions: Other: compare data patterns by data-driven algorithms to determine sepsis; Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality
- patients without pneumonia or sepsis (controls): Controls: Clinical phenotype of inflammation not due to suspected sepsis; patients with fever >38°C, C reactive Protein (CRP) >100mg/L, no infection focus expected in ≥ 24h.
  Interventions: Other: compare data patterns by data-driven algorithms to determine sepsis; Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality

INTERVENTIONS:
Other: compare data patterns by data-driven algorithms to determine sepsis — compare data patterns by data-driven algorithms including machine learning and multi-dimensional modelling to reliably determine sepsis
Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality — compare data patterns by data-driven algorithms including machine learning and multi-dimensional modelling to to predict sepsis-related mortality

SUMMARY:
This multi-center observational case-control study in Intensive Care Unit (ICU) patients is to identify novel biomarkers allowing to recognize severe community acquired pneumonia (sCAP) -associated sepsis at an earlier stage and predict sepsis-related mortality. Patients with sCAP (cases) will be profoundly characterized over time regarding the development of sepsis and compared with control patients. The mechanisms and influencing factors on the clinical course will be explored with most modern -omics technologies allowing a detailed characterisation. These data will be analysed using machine learning algorithms and multi-dimensional mathematical models.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU of one of the participating centers.
* Cases: severe community acquired pneumonia with requirement for ICU admission.
* Controls: Clinical phenotype of inflammation not due to suspected sepsis In addition, control patients will be patients with fever >38°C, CRP >100mg/L, no infection focus expected in ≥ 24h.
* All required sample types can most likely be collected within the first 24h visits.
* Expected ICU stay of more than 24h.

Exclusion Criteria:

* Admission to the hospital within the prior 14 days.
* Patients with psychosis
* Evidence of a hospital acquired pneumonia.
* One of the following respiratory conditions: Acute exacerbation of chronic obstructive pulmonary disease (COPD) or bronchiectasis, acute severe asthma, aspiration pneumonia, tuberculosis, clinical suspected viral pneumonia without bacterial infection, cardiogenic pulmonary oedema.
* Patients with an acute respiratory distress Syndrome (ARDS).
* Patient which can be managed as outpatients and do not require an ICU.
* Patient where a transmission to another institution is likely within the next 24h.
* Documented rejection of the general consent or participation to research in general.
* Patients with a palliative situation and a life expectancy due to other diseases (e.g. progressed cancer) less than 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients fulfilling the WHO-definition of a severe community acquired pneumonia (sCAP, cases) and patients with an inflammatory phenotype (controls) requiring intensive care medicine.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Detection of sepsis | within 7 days after study inclusion
  Sepsis detection based on new discovered digital biomarkers will be compared to classical sepsis-3 criteria (with an increase of the sequential organ failure assessment (SOFA) score of 2 or larger score points).
Sepsis related mortality | within 7 days after study inclusion
  Prediction of sepsis related mortality (with >80% sensitivity and specificity at least 24h prior to event)
Time to sepsis detection (minutes after Intensive Care Unit (ICU) admission) | within 7 days after study inclusion
  Time to sepsis detection (minutes after ICU admission) based on machine learning

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr., Principal Investigator — Clinical Microbiology, University Hospital Basel
Locations (15):
- Switzerland (15):
  - Clinical Bacteriology and Mycology, University Hospital Basel, Basel
  - Infectious Diseases and Hospital Epidemiology, University Hospital Basel, Basel
  - Intensive Care Unit; University Hospital Basel, Basel
  - Institute for Infectious Diseases, University of Bern, Bern
  - Infectious Diseases and Hospital Epidemiology, University Hospital Bern, Bern
  - Intensive Care Unit, University Hospital Bern, Bern
  - Clinical Bacteriology, University Hospital Geneva, Geneva
  - Infectious Diseases and Hospital Epidemiology, University Hospital Geneva, Geneva
  - Intensive Care Unit, University Hospital Geneva, Geneva
  - Clinical Microbiology, University Hospital Lausanne, Lausanne
  - Infectious Diseases and Hospital Epidemiology , University Hospital Lausanne, Lausanne
  - Intensive Care Unit, University Hospital Lausanne, Lausanne
  - Infectious Diseases and Hospital Epidemiology, University Hospital Zurich, Zurich
  - Institute for Medical Microbiology, University Hospital Zurich, Zurich
  - Intensive Care Unit, University Hospital Zurich, Zurich